CLINICAL TRIAL: NCT06465524
Title: Effects of High-Intensity Laser Therapy and Stretching Exercises on Chronic Non-Specific Neck Pain: Findings From a Clinical Trial
Brief Title: High-intensity Laser Therapy and Stretching Exercises for Chronic Non-specific Neck Pain: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quiropraxia y Equilibrio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13062024
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Non-specific Neck Pain
Keywords: Laser therapy; High-intensity laser therapy; Chronic pain; Neck pain; Clinical Trial
MeSH Terms: conditions — Chronic Pain; Neck Pain | interventions — Laser Therapy; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Experimental design of a double-blind, non-controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-intensity laser therapy and stretching exercise (Experimental): The BTL-6000 device, with 12W power and a wavelength of 1,064 nm, will administer laser therapy to the experimental group using the De la Barra et al. protocol. Treatment includes three phases: (Phase 1) Manual scanning 1: 12 W for 42 seconds, delivering 500 J over 100 cm2 per upper trapezius muscle (total 1,000 J). (Phase 2) Point technique: 4 W for 10 seconds per point (10 J per point), totaling 60 J per side (120 J total). (Phase 3) Manual scanning 2: 6 W for 83 seconds, delivering 500 J over 100 cm2 per upper trapezius muscle (total 1,000 J). Following the HILT treatment, we will perform three sets of 30 seconds each of passive bilateral static stretching exercises for the upper trapezius, levator scapulae, and scalene muscles.
  Interventions: Device: High-intensity laser therapy

INTERVENTIONS:
Device: High-intensity laser therapy — High-intensity laser therapy (HILT), also referred to as Class IV laser therapy, involves the administration of collimated and monochromatic electromagnetic radiation within the infrared or red spectrum. It operates at power levels exceeding 500 milliwatts (0.5 W), leveraging both photobiomodulation and thermal effects. This distinguishes HILT from Class III lasers (low-level laser therapy, or LLLT), which lack photothermal effects when operating below 500 mW.
  Other Names: Laser therapy; Power laser; Laser class IV

SUMMARY:
Chronic non-specific neck pain (CNNP) poses a significant challenge in healthcare, sparking interest in conservative and innovative therapeutic options such as high-intensity laser therapy (HILT). While evidence of its efficacy in this specific context remains limited, there is a robust foundation supporting the use of HILT in managing chronic neck pain, demonstrating effectiveness in pain reduction and functional improvement. Therefore, the aim of this study is to evaluate the clinical response to HILT treatment in patients with CNNP, investigating its potential therapeutic benefits and adverse effects. The findings of this study will provide valuable insights into the clinical experience with HILT in this population, serving as a pivotal starting point for future research in this field.

In a clinical trial, patients with CNNP will undergo a treatment regimen consisting of two weekly sessions of HILT and stretching exercises over four weeks. The study aims to assess primary outcomes such as resting pain intensity (RPI), movement pain intensity (MPI), and pain pressure threshold (PPT), measured using the numerical pain rating scale and algometry. Secondary outcomes will include cervical range of motion (CROM) and neck disability, assessed through inclinometry and the Neck Disability Index (NDI). Evaluations will occur post-treatment, with a follow-up assessment scheduled one month later.

DETAILED DESCRIPTION:
1.1 Study Type and Design: Experimental design for a non-controlled clinical trial.The study will be conducted in the Electrophysical Agents Laboratory (KIN 401) at the School of Physical Therapy, Faculty of Rehabilitation Sciences, Casona de las Condes Campus, Universidad Andrés Bello, located at Calle Fernández Concha Nº700, Las Condes, Santiago, Chile. The sample will be selected from the university population of the same faculty. The study group will be determined through a non-probabilistic sampling process. Participants will be recruited via a closed-ended questionnaire constructed according to selection criteria. The minimum number of participants required for the study will be calculated using the G-Power program, with a minimum of 20 participants. Subjects with CNNP pain will be recruited and will receive 8 sessions of HILT and stretching exercises over 4 weeks. Relevant outcomes will include resting pain intensity (RPI), movement pain intensity (MPI), and pressure pain threshold (PPT). Additionally, cervical range of motion (CROM) and neck disability (ND) will be assessed. Evaluations will be conducted at three time points: before treatment, at the end of treatment, and at a one-month follow-up evaluation.

1.2 Overall Objective To evaluate the effect of high-intensity laser therapy on reducing pain, increasing pain pressure threshold, improving cervical range of motion, and decreasing cervical disability in patients with non-specific chronic neck pain.

1.3 Specific Objectives - Determine the difference in cervical pain intensity before and after high-intensity laser therapy treatment.

* Assess the change in cervical pain pressure threshold before and after treatment with high-intensity laser therapy.
* Measure improvement in cervical range of motion in terms of flexion, extension, rotation, and lateral bending following high-intensity laser therapy.
* Evaluate the reduction in cervical disability using the cervical disability index before and after treatment with high-intensity laser therapy.
* Investigate the correlation between pain reduction, pain pressure threshold, improvement in range of motion, and reduction in cervical disability in response to high-intensity laser therapy.

1.4 Phases of the clinical trial

* Study Preparation and Design: In this initial stage, the experimental design of the non-controlled clinical trial will be established, defining study objectives and selecting key variables for measurement. Additionally, the laboratory environment will be prepared, and the research protocol will be designed.
* Treatment Implementation and Execution: During this phase, the study will be implemented, involving sample selection through a non-probabilistic sampling process, administration of the treatment (HILT and stretching exercises) to recruited participants, and collection of relevant clinical data.
* Evaluation and Results Analysis: The final stage will focus on evaluating the obtained results, including measurement of variables such as pain intensity, pain pressure threshold, cervical range of motion, and cervical disability. Statistical analyses will be conducted to determine treatment efficacy, and conclusions will be drawn based on the study findings.

2.1 Conceptual Definition of Variables:

- Pain intensity at rest: discomfort or more intense forms of pain localized in the cervical region, lateral neck, shoulders, or scapular region, reported by participants while at rest.

* Pain intensity at movement: discomfort or more intense forms of pain localized in the cervical region, lateral neck, shoulders, or scapular region, manifested by participants during neck movements.
* Pain pressure threshold: the minimum amount of pressure applied to a specific area of the body that induces the sensation of pain.
* Cervical range of motion: capacity of movement in the cervical spine, including movements in various anatomical planes such as flexion, extension, lateral bending, and rotation.
* Neck disability: limitation or restriction in neck functional capacity, manifested as difficulty in performing daily activities such as neck movement, maintaining an upright posture, performing work tasks, or engaging in recreational activities.
* Stretching exercises: static passive stretching exercises performed bilaterally by the therapist on the upper trapezius, levator scapulae, and scalene muscles, each held for 30 seconds with 30-second intervals, totaling 3 sets for each muscle group.
* High-intensity laser therapy uses concentrated laser light with power greater than 0.5 watts to treat musculoskeletal injuries, chronic pain, and promote healing through thermal effects and photobiomodulation.

2.2 Operational Definition of Variables: - Pain intensity at rest: assessed using the Numeric Pain Rating Scale (NPRS) from Gymna (R). measured on a scale from 0 to 10, where 0 represents no pain and 10 represents the most pain the participant reported.

- Pain intensity at movement: assessed using the Numeric Pain Rating Scale (NPRS) from Gymna (R). measured on a scale from 0 to 10, where 0 represents no pain and 10 represents the most pain the participant reported.

- Pain pressure threshold: assessed using pressure algometry with the FPX Wagner pressure algometer (R). The pressure threshold will be measured in pounds per square centimeter (lb/cm2).

- Cervical range of motion: assessed using inclinometry with the CROM device. The range of motion will be quantified in degrees (°).

- Neck disability is assessed using the Neck Disability Index (NDI). Cervical disability will be expressed as a percentage, where 0% indicates no disability and 100% indicates maximum disability.

* Stretching exercises: static and passive stretching exercises performed bilaterally by the therapist on the upper trapezius, levator scapulae, and scalene muscles. Each exercise will be held for 30 seconds with 30-second intervals, and 3 sets will be performed for each muscle group.
* High-intensity laser: application of a high-power laser using the BTL-6000 device at 12 Watts.

2.3 Types of Variables:

- Pain intensity at rest: dependent variable, ordinal qualitative.

* Pain intensity at movement: dependent variable, ordinal qualitative.
* Pain pressure threshold: dependent variable, continuous quantitative.
* Cervical range of motion: dependent variable, continuous quantitative.
* Neck disability: dependent variable, continuous quantitative.
* Cervical stretching exercises: independent variable, nominal qualitative.
* High-intensity laser therapy: independent variable, continuous quantitative.

  3. Ethical Considerations: The study received approval from the Ethics Committee of the Metropolitan East Health Service of Santiago, Chile, on October 26, 2022, in accordance with the principles of the Declaration of Helsinki (approval number 20200234).

  4. Participants: Participants will be recruited from the community of Universidad Andrés Bello. The study will be advertised through official channels, including email distribution and publication on the institutional website. Additionally, communication channels such as emails, social media, and panels within the Physical Therapy Department will be utilized. Volunteers will be contacted via telephone or email to attend the Electrophysical Agents Laboratory at the Faculty of Rehabilitation Sciences.

  5. Sample size: The sample size will be determined using G-Power software, considering a power of 90% (1-β), a confidence level of 95%, a significance level of 5% (α), and an effect size of 0.6. Previous studies in individuals with CNP have shown differences in pain intensity, favoring HILT plus exercise over ultrasound plus exercise. Therefore, a minimum sample size of 17 participants will be established. To accommodate potential dropouts during the study or follow-up, an additional 15% will be added to the sample, resulting in a total of at least 20 participants.

  6. Intervention: Participants will form a study group receiving HILT as an intervention. Alongside laser therapy, they will undergo a regimen of passive bilateral static stretching exercises targeting the upper trapezius, levator scapulae, and scalene muscles, with each stretch held for 30 seconds per set. These stretching exercises will be conducted immediately following the HILT treatment. The interventions will take place twice weekly over a span of four weeks, totaling eight sessions. These interventions will occur twice a week for four weeks, totaling eight sessions. Each treatment will be administered by an independent therapist ensuring intervention blindness.
* High-intensity laser therapy. For laser therapy, the BTL-6000 device with 12W power and a wavelength of 1,064 nm will be used. The treatment protocol integrates manual scanning and point techniques following De la Barra et al. It consists of three phases: Phase 1, manual scanning with 12 W power for 42 seconds per upper trapezius muscle, delivering 1,000 J in total; Phase 2, point technique (static) using 4 W power for 10 seconds per point, delivering 120 J in total; Phase 3, manual scanning with 6 W power for 83 seconds per upper trapezius muscle, delivering 1,000 J in total.
* Stretching exercise. Participants will also undergo passive bilateral static stretching exercises targeting the upper trapezius, levator scapulae, and scalene muscles. A therapist will administer these exercises, lasting 30 seconds each with a 30-second rest between sets, following the HILT treatment.

  7. Outcomes of Interest: The primary outcome measures will include resting pain intensity (RPI), pain intensity during movement (MPI), both assessed using the Numerical Pain Rating Scale (NPRS), and pain pressure threshold (PPT), evaluated with algometry. Algometry will assess six bilateral points across the cervical region, shoulders, and interscapular region. Secondary outcomes will encompass cervical range of motion (CROM), evaluated using inclinometry, and cervical disability, assessed with the Neck Disability Index (NDI). Evaluations will occur at three time points: baseline (before treatment), immediately post-treatment, and four weeks post-treatment (follow-up assessment). Two independent evaluators will conduct the assessments to ensure blindness in the evaluation process: one will handle the algometry assessment and NPRS application, while the other will handle the CROM evaluation. Neck disability will be assessed using the self-administered NDI questionnaire.

  8. Statistical Analysis: Descriptive statistics such as means, standard deviations, medians, and interquartile ranges will be used to analyze the variables RPI, MPI, PPT, CROM, and ND, based on data distribution. Tables will be created with demographic data such as gender and body mass index. For inferential analysis, tests for normality and homoscedasticity, such as the Shapiro-Wilk test and Bartlett's test, respectively, will be employed. Depending on the results, parametric or non-parametric tests will be selected: a one-way ANOVA or Kruskal-Wallis test to evaluate differences between sessions. Post-hoc analyses will be conducted using Tukey's or Bonferroni's tests for multiple comparisons. The significance level will be set at 0.05, and data analysis will be performed using IBM Statistical Package for the Social Sciences (SPSS) software (version 26; SPSS Inc.; Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Both sexes
* Experiencing chronic neck pain: Defined as pain or discomfort in the cervical region between the upper nuchal line and the T1 spinous process or the shoulder girdle. Lasting at least three months
* Neck Disability Index (NDI) score of 5 or higher
* Pain intensity of at least three on the Numerical Pain Rating Scale (NPRS) at rest

Exclusion Criteria:

* Any musculoskeletal injuries sustained in the neck or shoulders within the past three months
* The presence of osteosynthesis materials in the vicinity of the shoulders, neck, or surrounding areas
* The existence of skin wounds or changes, such as psoriasis, scars, or burns, in the neck or shoulder region.
* Continuous usage of analgesic medication, anti-inflammatories, or muscle relaxants.
* Neurological disorders, which include paresthesias, partial or total loss of sensation, decreased strength, and color changes in the neck, arms, forearms, or hands.
* Diagnosis of photosensitivity
* Skin types V and VI, as determined by the Fitzpatrick scale
* Solar urticaria or adverse reactions to sunlight are present.
* Diagnosis of autoimmune diseases (e.g., dermatomyositis, systemic lupus erythematosus, hepatic porphyria, carcinoid syndrome, pellagra)
* Diagnosis of cancer or tumors within the past five years
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity at rest (numeric pain rating scale, NPRS) | Baseline, 4 weeks (8 sessions) and 4 weeks (follow-up)
  Magnitude of neck pain reported by participants at rest. The pain intensity at rest will be measured with the numeric pain rating scale (NPRS). The scale quantifies pain from 0 to 10, where 0 represents the absence of pain and 10 represents the maximum tolerable pain.
Pain intensity at movement (numeric pain rating scale, NPRS) | Baseline, 4 weeks (8 sessions) and 4 weeks (follow-up)
  Magnitude of pain reported by participants during active cervical movements, including flexion, extension, lateral bending, and rotation. The pain intensity during movement will be measured with the numeric pain rating scale (NPRS).The scale quantifies pain from 0 to 10, where 0 represents the absence of pain and 10 represents the maximum tolerable pain.
Pain pressure threshold (algometry) | Baseline, 4 weeks (8 sessions) and 4 weeks (follow-up)
  The maximum mechanical pressure tolerated by the patient was assessed using algometry. Six bilateral points were evaluated: 2 cm lateral to the spinous processes of C2, C5, T4, and T8; the midpoint of the upper trapezius muscle (between C7 and the acromion); the levator scapulae (2 cm superior to the superior angle of the scapula); and the middle third of the right tibialis anterior muscle. The pain pressure threshold will be evaluated with pressure algometry (FPX Wagner (R) equipment). The pain pressure threshold measurement unit will be evaluated in pounds per square centimeter.

SECONDARY OUTCOMES:
Cervical range of movement (inclinometer) | Baseline, 4 weeks (8 sessions) and 4 weeks (follow-up)
  The cervical range of motion refers to the extent of movement achievable by the cervical spine in various directions, including flexion (forward bending), extension (backward bending), lateral flexion (side bending to the left and right), and rotation (turning left and right). The cervical range of motion will be assessed using an inclinometry device (CROM device). The degrees of movement are quantified for each active osteokinematic movement performed by the participant.
Neck disability (neck disability index) | Baseline, 4 weeks (8 sessions) and 4 weeks (follow-up)
  Neck disability refers to the extent or degree to which cervical pain and associated symptoms impact a person's ability to perform daily activities and participate in normal life roles. It will be assessed using the Neck Disability Index (NDI), which will evaluate the functional limitations and subjective experiences related to neck pain and its effects on a person's quality of life. Cervical disability will be quantified as a percentage (0% absence of disability and 100% maximum disability reported by the participant).

CONTACTS AND LOCATIONS:
Overall Officials: Hernán Andrés de la Barra Ortiz, PhD(c), Principal Investigator — Andrés Bello University
Locations (1):
- Universidad Andrés Bello, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data (IPD) available to other researchers. There is an intention to publish the study protocol.

REFERENCES:
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Mayoral-Del-Moral O, Pacheco-da-Costa S, Prieto-Merino D, Sanchez-Sanchez B. Health related quality of life improvement in chronic non-specific neck pain: secondary analysis from a single blinded, randomized clinical trial. Health Qual Life Outcomes. 2018 Nov 6;16(1):207. doi: 10.1186/s12955-018-1032-6. PMID 30400984
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Mayoral-Del Moral O, Sanchez-Sanchez B, Dommerholt J, Gutierrez-Ortega C. Prevalence of Myofascial Pain Syndrome in Chronic Non-Specific Neck Pain: A Population-Based Cross-Sectional Descriptive Study. Pain Med. 2016 Dec;17(12):2369-2377. doi: 10.1093/pm/pnw114. Epub 2016 Jun 20. PMID 28025371
- [Background] Ortego G, Villafane JH, Domenech-Garcia V, Berjano P, Bertozzi L, Herrero P. Is there a relationship between psychological stress or anxiety and chronic nonspecific neck-arm pain in adults? A systematic review and meta-analysis. J Psychosom Res. 2016 Nov;90:70-81. doi: 10.1016/j.jpsychores.2016.09.006. Epub 2016 Sep 9. PMID 27772562
- [Background] Opara M, Kozinc Z. Which muscles exhibit increased stiffness in people with chronic neck pain? A systematic review with meta-analysis. Front Sports Act Living. 2023 Aug 30;5:1172514. doi: 10.3389/fspor.2023.1172514. eCollection 2023. PMID 37712006
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399
- [Background] Castellini G, Pillastrini P, Vanti C, Bargeri S, Giagio S, Bordignon E, Fasciani F, Marzioni F, Innocenti T, Chiarotto A, Gianola S, Bertozzi L. Some conservative interventions are more effective than others for people with chronic non-specific neck pain: a systematic review and network meta-analysis. J Physiother. 2022 Oct;68(4):244-254. doi: 10.1016/j.jphys.2022.09.007. Epub 2022 Oct 17. PMID 36266185
- [Background] Huang JF, Meng Z, Zheng XQ, Qin Z, Sun XL, Zhang K, Tian HJ, Wang XB, Gao Z, Li YM, Wu AM. Real-World Evidence in Prescription Medication Use Among U.S. Adults with Neck Pain. Pain Ther. 2020 Dec;9(2):637-655. doi: 10.1007/s40122-020-00193-1. Epub 2020 Sep 17. PMID 32940899
- [Background] Fredin K, Loras H. Manual therapy, exercise therapy or combined treatment in the management of adult neck pain - A systematic review and meta-analysis. Musculoskelet Sci Pract. 2017 Oct;31:62-71. doi: 10.1016/j.msksp.2017.07.005. Epub 2017 Jul 21. PMID 28750310
- [Background] Martimbianco ALC, Porfirio GJ, Pacheco RL, Torloni MR, Riera R. Transcutaneous electrical nerve stimulation (TENS) for chronic neck pain. Cochrane Database Syst Rev. 2019 Dec 12;12(12):CD011927. doi: 10.1002/14651858.CD011927.pub2. PMID 31830313
- [Background] Hakkinen A, Salo P, Tarvainen U, Wiren K, Ylinen J. Effect of manual therapy and stretching on neck muscle strength and mobility in chronic neck pain. J Rehabil Med. 2007 Sep;39(7):575-9. doi: 10.2340/16501977-0094. PMID 17724558
- [Background] Chow R. EBM in action: is laser treatment effective and safe for musculoskeletal pain? Med J Aust. 2002 Feb 18;176(4):194-5. doi: 10.5694/j.1326-5377.2002.tb04366.x. No abstract available. PMID 11913929
- [Background] de la Barra Ortiz HA, Arias M, Liebano RE. A systematic review and meta-analysis of randomized controlled trials on the effectiveness of high-intensity laser therapy in the management of neck pain. Lasers Med Sci. 2024 May 6;39(1):124. doi: 10.1007/s10103-024-04069-0. PMID 38709332
- [Background] Clijsen R, Brunner A, Barbero M, Clarys P, Taeymans J. Effects of low-level laser therapy on pain in patients with musculoskeletal disorders: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2017 Aug;53(4):603-610. doi: 10.23736/S1973-9087.17.04432-X. Epub 2017 Jan 30. PMID 28145397
- [Background] Chow RT, David MA, Armati PJ. 830 nm laser irradiation induces varicosity formation, reduces mitochondrial membrane potential and blocks fast axonal flow in small and medium diameter rat dorsal root ganglion neurons: implications for the analgesic effects of 830 nm laser. J Peripher Nerv Syst. 2007 Mar;12(1):28-39. doi: 10.1111/j.1529-8027.2007.00114.x. PMID 17374099
- [Background] Cotler HB, Chow RT, Hamblin MR, Carroll J. The Use of Low Level Laser Therapy (LLLT) For Musculoskeletal Pain. MOJ Orthop Rheumatol. 2015;2(5):00068. doi: 10.15406/mojor.2015.02.00068. Epub 2015 Jun 9. PMID 26858986
- [Background] de la Barra Ortiz HA, Avila MA, Miranda LG, Liebano RE. Effect of high-intensity laser therapy in patients with non-specific chronic neck pain: study protocol for a randomized controlled trial. Trials. 2023 Aug 31;24(1):563. doi: 10.1186/s13063-023-07599-0. PMID 37653525
- [Background] Arroyo-Fernandez R, Aceituno-Gomez J, Serrano-Munoz D, Avendano-Coy J. High-Intensity Laser Therapy for Musculoskeletal Disorders: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. J Clin Med. 2023 Feb 13;12(4):1479. doi: 10.3390/jcm12041479. PMID 36836014
- [Background] Chow RT, Johnson MI, Lopes-Martins RA, Bjordal JM. Efficacy of low-level laser therapy in the management of neck pain: a systematic review and meta-analysis of randomised placebo or active-treatment controlled trials. Lancet. 2009 Dec 5;374(9705):1897-908. doi: 10.1016/S0140-6736(09)61522-1. Epub 2009 Nov 13. PMID 19913903
- [Background] Shrestha B, Dunn L. The Declaration of Helsinki on Medical Research involving Human Subjects: A Review of Seventh Revision. J Nepal Health Res Counc. 2020 Jan 21;17(4):548-552. doi: 10.33314/jnhrc.v17i4.1042. PMID 32001865
- [Background] Proehl JA, Alexander S, Manton AP. Integrity and Transparency in Reporting Clinical Trials. Adv Emerg Nurs J. 2017 Jan/Mar;39(1):1-2. doi: 10.1097/TME.0000000000000136. No abstract available. PMID 28141604
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Andrade C. Sample Size and its Importance in Research. Indian J Psychol Med. 2020 Jan 6;42(1):102-103. doi: 10.4103/IJPSYM.IJPSYM_504_19. eCollection 2020 Jan-Feb. PMID 31997873
- [Background] Dundar U, Turkmen U, Toktas H, Solak O, Ulasli AM. Effect of high-intensity laser therapy in the management of myofascial pain syndrome of the trapezius: a double-blind, placebo-controlled study. Lasers Med Sci. 2015 Jan;30(1):325-32. doi: 10.1007/s10103-014-1671-8. Epub 2014 Oct 2. PMID 25274197
- [Background] Page P. Current concepts in muscle stretching for exercise and rehabilitation. Int J Sports Phys Ther. 2012 Feb;7(1):109-19. PMID 22319684
- [Background] Tunwattanapong P, Kongkasuwan R, Kuptniratsaikul V. The effectiveness of a neck and shoulder stretching exercise program among office workers with neck pain: a randomized controlled trial. Clin Rehabil. 2016 Jan;30(1):64-72. doi: 10.1177/0269215515575747. Epub 2015 Mar 16. PMID 25780258
- [Background] Rampazo EP, de Andrade ALM, da Silva VR, Back CGN, Liebano RE. Photobiomodulation therapy and transcutaneous electrical nerve stimulation on chronic neck pain patients: Study protocol clinical trial (SPIRIT Compliant). Medicine (Baltimore). 2020 Feb;99(8):e19191. doi: 10.1097/MD.0000000000019191. PMID 32080103
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Rampazo da Silva EP, Silva VR, Bernardes AS, Matuzawa F, Liebano RE. Segmental and extrasegmental hypoalgesic effects of low-frequency pulsed current and modulated kilohertz-frequency currents in healthy subjects: randomized clinical trial. Physiother Theory Pract. 2021 Aug;37(8):916-925. doi: 10.1080/09593985.2019.1650857. Epub 2019 Aug 12. PMID 31402740
- [Background] Williams MA, McCarthy CJ, Chorti A, Cooke MW, Gates S. A systematic review of reliability and validity studies of methods for measuring active and passive cervical range of motion. J Manipulative Physiol Ther. 2010 Feb;33(2):138-55. doi: 10.1016/j.jmpt.2009.12.009. PMID 20170780
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Andrade Ortega JA, Delgado Martinez AD, Almecija Ruiz R. Validation of the Spanish version of the Neck Disability Index. Spine (Phila Pa 1976). 2010 Feb 15;35(4):E114-8. doi: 10.1097/BRS.0b013e3181afea5d. PMID 20110848
- [Background] MacDermid JC, Walton DM, Avery S, Blanchard A, Etruw E, McAlpine C, Goldsmith CH. Measurement properties of the neck disability index: a systematic review. J Orthop Sports Phys Ther. 2009 May;39(5):400-17. doi: 10.2519/jospt.2009.2930. PMID 19521015
- [Background] Mishra P, Pandey CM, Singh U, Gupta A, Sahu C, Keshri A. Descriptive statistics and normality tests for statistical data. Ann Card Anaesth. 2019 Jan-Mar;22(1):67-72. doi: 10.4103/aca.ACA_157_18. PMID 30648682
- See also: A Randomized Comparative Study between High-Intensity Laser Therapy and Ultrasound Therapy on Chronic Neck Pain among Adult Patients — http://dspace.alquds.edu/handle/20.500.12213/7597